CLINICAL TRIAL: NCT01123525
Title: Adenosine Instead of Supranormal Potassium in Crystalloid Cardioplegia, a Randomized Clinical Study
Brief Title: Adenosine Cardioplegia; Improved Cardioprotection?
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AdCard 2010; 2008-004274-40 (EudraCT Number)
Record Dates: First submitted 2010-04-30; First posted 2010-05-14 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Angina Pectoris
MeSH Terms: conditions — Angina Pectoris | interventions — Adenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Adenosine cardioplegia (Experimental): Adenosine cardioplegia
  Interventions: Drug: Adenosine
- Control (Active Comparator): Standard hyperkalemic cardioplegia
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Adenosine — 1.2 mM adenosine instead of supranormal potassium in the cardioplegic solution

SUMMARY:
60 elective patients for CABG will be included to receive either standard hyperkalemic cardioplegia (St.Thomas Hospital Solution No I) or cardioplegia where supranormal potassium is replaced with 1.2 mM adenosine. Hypothesis as follows: 1. Adenosine instead of supranormal potassium in the cardioplegic solution give satisfactory cardiac arrest. 2. Adenosine instead of supranormal potassium in the cardioplegic solution gives equal cardioprotection. The patients will be followed with PiCCO-catheter to monitor cardiac function and repetitive blood samples to measure release of cardiac enzymes.

ELIGIBILITY:
Inclusion Criteria:

* Elective patients
* Ejection fraction > 40%
* Age 40-75
* No release og TnT or CKMB within last week before CABG
* Pure CABG

Exclusion Criteria:

* Age >75 or < 40
* EF < 40%
* Emergency operations
* Unstable angina
* Release of TnT or CKMB within the week before operation

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Release of cardiac enzymes (TnT and CKMB) | First 48 hour postoperatively
  Repeatedly measured postoperatively.

SECONDARY OUTCOMES:
PiCCO | First 24 hours postoperatively
  Measurement of cardiac function and hemodynamics the first 24 hours postoperatively
Endothelial injury | Peroperatively (before crossclamping aorta and after 5 minutes of reperfusion)
  Measurements of markers of endothelial injury/dysfunction peroperatively. Blood will be sampled immediately before cross-clamping the aorta and after 5 minutes of reperfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of North Norway, Troomsø, Norway

REFERENCES:
- [Derived] Jakobsen O, Naesheim T, Aas KN, Sorlie D, Steensrud T. Adenosine instead of supranormal potassium in cardioplegia: it is safe, efficient, and reduces the incidence of postoperative atrial fibrillation. A randomized clinical trial. J Thorac Cardiovasc Surg. 2013 Mar;145(3):812-8. doi: 10.1016/j.jtcvs.2012.07.058. Epub 2012 Sep 7. PMID 22964356